CLINICAL TRIAL: NCT02911220
Title: Genetic Study of Familial Forms of Non-atopic Asthma
Acronym: GANA
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: not enough available families to get significant genetic results
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: RC15_0354; 2016-A00922-49 (Other: ANSM)
Record Dates: First submitted 2016-09-09; First posted 2016-09-22 (Estimated); Last update posted 2021-01-20 (Actual); Status verified 2021-01

CONDITIONS: Non-atopic Asthma; Genetic Study

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- blood sample for genetic evaluation (Other): a blood sample is collected once for genetic analysis
  Interventions: Genetic: demonstration of genetic mutations causing non-atopic asthma

INTERVENTIONS:
Genetic: demonstration of genetic mutations causing non-atopic asthma — recruitment of familial forms of non-atopic asthma (patients with non-atopic asthma and their relatives) to perform genetic analysis of exome sequencing

SUMMARY:
The intrinsic asthma (atopic or not) is a particular phenotype marked by an early later symptoms, increased severity, sensitivity associated with nonsteroidal anti-inflammatory drugs (NSAIDs), a sinonasal polyposis and eosinophilia.

Unlike allergic asthma, this form does not today demonstrated its genetic character. However, the existence of familial forms of asthma in this region Pays de La Loire led us to hypothesize the existence of genetic variations can explain some familial forms of non-atopic asthma. Corresponding genes may be relevant to understanding the pathophysiological pathways involved in the more common sporadic forms.

The investigators propose a study combining genetic linkage analysis and complete sequencing exomes to identify one or more genetic abnormalities associated with non-atopic asthma. The clinical stage essential for mutation identification is to identify and recruit large families with members affected by non-atopic asthma and ensure accurate phenotyping of all individuals recruited over several generations.

The aim of this study is to create a cohort of families who have more members within them non-atopic asthma. A high genetic combined exome sequencing throughput analysis in a family linkage study will then reveal the presence or absence of genetic variations associated with intrinsic asthma.

DETAILED DESCRIPTION:
Patients with non-atopic asthma will be identified in consultation pulmonology at Laennec Hospital (CHU Nantes) from the consultant population to severe asthma.

These patients will be treated as index case.

The investigator will conduct a family tree of the index case to identify families where the number of healthy individuals and those with non-atopic asthma makes relevant a family genetic study. Before initiating the family screening, it is necessary to have notion of at least two individuals carrying non-atopic asthma at least two generations in the family.

Related agreeing to participate in this study will be included.

ELIGIBILITY:
Inclusion Criteria:

* index case:

  * Major
  * Lack of respiratory disease documented in the medical record other than asthma
  * Severe Asthma by definition ATS / ERS 2014:
* Treatment with high doses of CI and beta2 agonists for long-acting (B2LDA) or anti leukotriene or theophylline during the previous year or oral corticosteroids (CO) more than 50% from the previous year to prevent loss of control asthma.
* Asthma "uncontrolled" (at least 1 criteria):

  * ACT <20 and / or ACQ> 1.5 (Asthma Control Test)
  * 2 courses or more CO in the previous year
  * 1 hospitalization for asthma in the previous year
  * FEV <80% predicted despite bronchodilators.
* Examination or medical record to find at least one member of the genetically non-atopic asthma associated family
* Prick negative tests for common allergens, questionnaire seeking negative atopy (SFAR Love) Phadiatop or negative diagnosis of non-atopic asthma confirmed by the adjudication committee
* informed and written consent of the patient to participate in the study
* Affiliated to a social security scheme

Exclusion Criteria:

* Pregnant women
* Minors

  - Known associated respiratory pathologies (COPD, bronchial dilatation, diffuse infiltrating pneumopathy)
* Major Trust
* Subject having demonstrated the inability or refusal to sign an informed consent

Relatives' patients:

* Major
* Related to the 1st and 2nd level of the index case or another member with family
* Related with or without a asthma (atopic or non-atopic)
* Informed and written consent of the patient to participate in the study Affiliated to a social security scheme

Exclusion Criteria:

* Pregnant women
* Minors
* Major Trust
* Subject having demonstrated the inability or refusal to sign an informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2020-02-26 (Actual); Primary Completion 2020-02-26 (Actual); Study Completion 2020-02-26 (Actual)

PRIMARY OUTCOMES:
broadband genetic and fine characterization of the phenotype in familial forms. | 36 months

SECONDARY OUTCOMES:
Identification of a homogeneous group of non-atopic asthma patients | 36 months

CONTACTS AND LOCATIONS:
Locations (1):
- CHU de Nantes - Service de Pneumologie - HGRL, Nantes, France